CLINICAL TRIAL: NCT00597285
Title: HHV6B in Epilepsy Imaging and CSF Studies
Brief Title: Relationship of HHV-6B Virus to Seizures and Brain Injury
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080027; 08-N-0027
Record Dates: First submitted 2008-01-08; First posted 2008-01-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2013-11-01

CONDITIONS: Epilepsy; HHV6B Infection
Keywords: 18-F-Fluoro-2-Deoxy-D-Glucose (FDG); Magnetic Resonance; Epilepsy; HHV-6B; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will look for evidence that a virus called HHV-6B may be related to seizures and to a form of brain injury called mesial temporal sclerosis that is associated with seizures. The study will use new, more sensitive brain scans to try to detect brain regions that might be affected by the virus and will examine cerebrospinal fluid (CSF, the fluid that bathes the brain and spinal cord) for evidence of the virus as well.

Healthy volunteers and people with seizures uncontrolled by anti-epileptic drugs who are between 18 and 45 years of age may be eligible for this study. Candidates are screened with a physical examination and laboratory tests.

Participants undergo the following procedures:

* PET scan. This test uses a radioactive chemical called 18FDG, which is detected by the PET scanner to obtain images of the brain. The subject lies on a table with his or her head positioned in the scanner. A swimming cap with a small light reflector is placed on the head to monitor the position of the head during the scan. A catheter (plastic tube) is inserted into an artery at the wrist or elbow crease of the arm for obtaining blood samples during the scan, and a second catheter is placed in a vein in the other arm for injecting the 18FDG. The scan takes up to 2 hours. A second scan may be done over an additional 15 minutes.
* MRI. This test uses a strong magnetic field and radio waves to obtain images of the brain. The subject lies on a table that can slide in and out of a metal cylinder surrounded by a magnetic field. Most scans last between 45 and 90 minutes.
* Lumbar puncture. The subject sits upright or lies on a table with the knees curled to the chest for this procedure. A local anesthetic is injected to numb the skin and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Blood tests. About 4 tablespoons of blood are drawn for viral tests.

DETAILED DESCRIPTION:
Objectives: 1) to attempt to detect specific patterns of hippocampal injury in patients with temporal lobe epilepsy that may be associated with HHV-6B infection; 2) To attempt to detect evidence for persistent HHV6 infection in CSF in patients with refractory temporal lobe epilepsy. 3) to obtain preliminary pilot data on the ability of high resolution structural to detect abnormalities in epilepsy patients not seen with standard scanners.

Study Population: 45 patients with localization-related epilepsy; 45 healthy volunteers

Design: 1) imaging with a 7T MRI magnetic resonance scanner; 2) Lumbar puncture. 3) blood sampling

Main outcome measure: 1) Detection of evidence for HHV6 infection in CSF

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be avaluated for participation under screening protocol 01-N-0139.

Patients

Male and female subjects age 18 to 55

Subjects with seizures uncontrolled by antiepileptic drugs

Subjects with no other illnesses, or taking other substances or medicines that could interfere with the study

Healthy Controls

Male and female subjects age 18 to 55.

EXCLUSION CRITERIA:

Patient

Subjects who are pregnant or breast feeding.

Subjects with any medical condition that could interfere with the study.

Subjects who are taking drugs that significantly reduce blood clotting such as Coumadin or Warfarin.

Healthy Volunteers

Subjects who are pregnant or breast feeding

Subjects who have any medical condition or be taking any substance or medication that could interfere with the study

Subjects who are taking drugs that significantly reduce blood cloting such as Coumadin or Warfarin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-01-03; Study Completion 2013-11-01

PRIMARY OUTCOMES:
Detection of evidence for HHV6 infection in CSF

SECONDARY OUTCOMES:
Detection of lesions on 7T compared to 3T MRI

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker GA, Nashef L, van Hout BA. Current issues in the management of epilepsy: the impact of frequent seizures on cost of illness, quality of life, and mortality. Epilepsia. 1997;38 Suppl 1:S1-8. doi: 10.1111/j.1528-1157.1997.tb04511.x. PMID 9092951
- [Background] Begley CE, Famulari M, Annegers JF, Lairson DR, Reynolds TF, Coan S, Dubinsky S, Newmark ME, Leibson C, So EL, Rocca WA. The cost of epilepsy in the United States: an estimate from population-based clinical and survey data. Epilepsia. 2000 Mar;41(3):342-51. doi: 10.1111/j.1528-1157.2000.tb00166.x. PMID 10714408
- [Background] Berg AT, Vickrey BG, Testa FM, Levy SR, Shinnar S, DiMario F, Smith S. How long does it take for epilepsy to become intractable? A prospective investigation. Ann Neurol. 2006 Jul;60(1):73-9. doi: 10.1002/ana.20852. PMID 16685695